CLINICAL TRIAL: NCT01803919
Title: Multicentric, Controlled, Randomized Clinical Trial to Assess the Efficacy and Cost-effectiveness of Urinary Catheters With Silver Alloy Coating Versus Conventional Catheters in Spinal Cord Injured Patients
Brief Title: Efficacy Study of Antimicrobial Catheters to Avoid Urinary Infections in Spinal Cord Injured Patients
Acronym: ESCALE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Asociacion Colaboracion Cochrane Iberoamericana (Other); European Clinical Research Infrastructure Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIBSP-SUR-2011-68; 112210 (Other Grant/Funding Number: La Fundació La Marató de TV3)
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Tract Infection
Keywords: Spinal cord injuries; Urinary tract infection; Urinary catheters; Protocol; Randomized clinical trial
MeSH Terms: conditions — Urinary Tract Infections; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silver Alloy-Coated Urinary Catheters (Experimental): Bactiguard® Infection Protection coating consists of noble metals such as gold, palladium and silver. Trained health staff performs urethral catheterization and select the most adequate catheter size. To ensure aseptic conditions they are asked to strictly follow the current protocol in their respective centers. Indwelling urethral catheters are periodically replaced about 30 days of use; to not interfere with current clinical practice, the policy of each center (or the investigator criteria) for catheter replacement and removal is considered valid for this study.
  Interventions: Device: Silver Alloy-Coated Urinary Catheters
- Conventional Urinary Catheter (Other): Conventional or standard urinary catheters are those commonly used in each study center, most of them made of silicone or silicone-latex. Trained health staff performs urethral catheterization and select the most adequate catheter size. To ensure aseptic conditions they are asked to strictly follow the current protocol in their respective centers. Indwelling urethral catheters are periodically replaced about 30 days of use; to not interfere with current clinical practice, the policy of each center (or the investigator criteria) for catheter replacement and removal is considered valid for this study.
  Interventions: Device: Conventional Urinary Catheter

INTERVENTIONS:
Device: Silver Alloy-Coated Urinary Catheters
  Other Names: BIP Foley catheter - Silicone Bactiguard Infection Protection
  Arms: Silver Alloy-Coated Urinary Catheters
Device: Conventional Urinary Catheter
  Other Names: Foley silicona 100% (16 or 18 Ch); Foley Rüsch (16 or 18 Ch); Foley Bardex (16 or 18 Ch); Folysil (16 or 18 Ch); Foley Rochester (16 or 18 Ch); Foley Euromedical (16 or 18 Ch)
  Arms: Conventional Urinary Catheter

SUMMARY:
The purpose of this trial is to make a comparison between the use of antiseptic silver alloy-coated silicone urinary catheters and the use of conventional silicone urinary catheters in spinal cord injured patients to prevent urinary infections.

DETAILED DESCRIPTION:
Antiseptic Silver Alloy-Coated Silicone Urinary Catheters seems to be a promising intervention to reduce urinary tract infections; however, research evidence cannot be extrapolated to spinal cord injured patients.

The study is an open, randomized, multicentric, and parallel clinical trial with blinded assessment. The study includes spinal cord injured patients who require at least seven days of urethral catheterization as a method of bladder voiding. Participants are on-line centrally randomized and allocated to one of the two interventions (Antiseptic Urinary Catheters or Conventional Catheters). Catheters are used for a maximum period of 30 days or removed earlier at the clinician criteria.

The main outcome is the incidence of urinary tract infections by the time of catheter removal or at day 30 after catheterization, the event that occurs first. Intention-to-treat analysis will be performed, as well as a primary analysis of all patients.

The aim of this study is to assess whether silver alloy-coated silicone urinary catheters reduce urinary infections in spinal cord injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with traumatic or medical spinal cord injury
* Age of 18 years or above
* Patients who need an indwelling urinary catheter as a method of bladder drainage for at least 7 days.
* Patients who are willing to participate in the study and give their written informed consent (If a patient is unable to give written consent because of physical or mental disability, an affirmation of consent will be taken in his presence from his relative or legal guardian).

Exclusion Criteria:

* Patients who can benefit from other method of bladder drainage such as intermittent catheterization, suprapubic drainage, reflex voiding or use of an external collector.
* Patients with urinary tract infection at the moment of inclusion
* Current antibiotic use or use within 7 days prior to inclusion
* Outpatients with sporadic medical examinations (less than one per month)
* Known allergy to latex, silver salts or hydrogels.
* Patients with surgical interventions in the urinary tract that may interfere, at the investigator criteria, with the study results.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter associated urinary tract infection | at any time from catheterization procedure and 30th day, catheter removal or catheter replacement (whichever occurs first)
  Is considered that a patient suffer a urinary tract infection if they have at least one suggestive sign or symptom with no other recognized cause and a positive urine culture with no more than 2 species of microorganisms.
  An urinary tract infection is considered catheter associated if the specimen collection is performed at any time from catheterization procedure and 30th day, catheter removal or catheter replacement (whichever occurs first).

SECONDARY OUTCOMES:
Asymptomatic urinary tract infection | at any time from catheterization procedure and 30th day, catheter removal or catheter replacement (whichever occurs first)
  A positive urine culture with no more than 2 species of microorganisms(collected at any time from catheterization procedure and 30th day, catheter removal or catheter replacement, whichever occurs first), and no signs or symptoms.
Bacteremic urinary tract infection | at any time from catheterization procedure and 30th day, catheter removal or catheter replacement (whichever occurs first)
  Those with the primary outcome and with a positive blood culture with at least 1 matching uropathogen microorganism to the urine culture.

OTHER OUTCOMES:
Direct costs | From catheterization procedure and 30th day, catheter removal or catheter replacement or finalization of complication(s) or related treatment(s), whichever last longer.
  Calculation of direct costs attributable to the use of intervention or control urinary catheters and their complications
Number of participants with adverse events related to catheterization as a Measure of Safety and Tolerability | at any time from catheterization procedure and 30th day, catheter removal or catheter replacement (whichever occurs first)
  Any untoward medical occurrence related to urinary catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bonfill, MD, PhD, Principal Investigator — Asociacion Colaboracion Cochrane Iberoamericana
Locations (20):
- Mutual de la Seguridad Chilena, Santiago, Chile
- Italy (4):
  - Azienda Ospedaliero-Universitaria - Ospedali Riuniti di Ancona - Unità Spinale, Ancona
  - Azienda Ospedaliero-Universitaria Policlinico di Bari- Unità Operativa di Medicina Fisica e Riabilitazione e Unità Spinale Unipolare, Bari
  - Unità Operative Recupero e Riabilitazione Funzionale e Gravi Cerebrolesioni Acquisite, Ceglie Messapica
  - Unità Spinale Unipolare, Rome
- Portugal (3):
  - Centro de Medicina de Reabilitação de Alcoitão, Alcoitão, Alcabideche
  - Centro Clínico Académico - Braga, Associação (2CA-Braga), Braga
  - Centro Hospitalar do Porto, Porto
- Spain (10):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital de Neurorrehabilitación Instituto Guttmann, Badalona, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz, Cadiz
  - Complejo Hospitalario Universitario Insular - Materno Infantil de Canarias, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Nacional de Parapléjicos, Toledo, Toledo
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
- Turkey (Türkiye) (2):
  - Dokuz Eylul University Dept. of Physical Medicine and Rehabilitation, Alsancak, İzmir
  - Ege University Dept. of Physical Medicine and Rehabilitation, Bornova, İzmir

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bonfill X, Rigau D, Jauregui-Abrisqueta ML, Barrera Chacon JM, de la Barrera SS, Aleman-Sanchez CM, Bea-Munoz M, Moraleda Perez S, Borau Duran A, Espinosa Quiros JR, Ledesma Romano L, Fuertes ME, Araya I, Martinez-Zapata MJ. A randomized controlled trial to assess the efficacy and cost-effectiveness of urinary catheters with silver alloy coating in spinal cord injured patients: trial protocol. BMC Urol. 2013 Jul 30;13:38. doi: 10.1186/1471-2490-13-38. PMID 23895463